CLINICAL TRIAL: NCT00768651
Title: Pilot Study of Safety and Efficacy of Combined Use of Dipeptidyl-peptidase Inhibitor (Sitagliptin) and Proton Pump Inhibitor (Pantoprazole) to Prevent Beta-cell Apoptosis and Promote Islet Regeneration in Islet Transplant Recipients With Early Graft Dysfunction
Brief Title: Incretin Effect and Use After Clinical Islet Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7331
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Results first posted 2015-06-18 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Pantoprazole; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- One arm: Sitagliptin + Pantoprazole (Experimental): Intervention Details:
  Sitagliptin 100 mg daily and Pantoprazole 40 mg bid for 6 months, followed by a three-month washout.
  Interventions: Drug: Pantoprazole; Drug: Sitagliptin

INTERVENTIONS:
Drug: Pantoprazole — Starting on Day 1, Pantoprazole 80 mg daily (40 mg every morning and 40 mg every evening) administered orally at the same time each day for a period of 6 months.
  Other Names: Pantoloc
Drug: Sitagliptin — Starting on Day 1, Sitagliptin 100mg once daily administered orally at the same time each day for a period of 6 months.
  Other Names: Januvia

SUMMARY:
We aim to study if the administration of medications to increase the secretion of hormones from the intestines can improve glycemic control, reduce insulin use and promote β-cell regeneration/expansion in subjects with type 1 diabetes following islet transplantation who are back using small doses of insulin because of early graft dysfunction. We believe that the results will enable us to understand whether these drugs could be useful in islet transplant recipients, particularly if glycemic control deteriorates.

DETAILED DESCRIPTION:
This is a single centre non-randomized pilot study. Subjects will be recruited from the current cohort of islet transplant recipients at the University of Alberta.

The primary objective of the study is to evaluate whether the combination of sitagliptin and pantoprazole can restore insulin independence in previously insulin independent islet transplant recipients experiencing early graft dysfunction. The study will also evaluate the safety of the combination drug therapy.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet the following criteria to be enrolled in this study:

1. Male or female, aged 18 to 70, inclusive, who is a previous islet transplant recipient (at least 3 months since last islet transplant) and who received their transplant at the University of Alberta.
2. Insulin independent for 3 months or longer after islet transplant.
3. Early graft dysfunction as defined by:

   1. HbA1c >6% (but less than 7.5%); or
   2. fasting glucose > 7 mmol/L (126 mg/dl); or
   3. random glucose > 10 mmol/L (180 mg/dl), and
   4. Total insulin use of < 10 units/day.
4. C-peptide positive.
5. Able to provide informed consent.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. Unable to provide informed consent.
2. Prior therapy with sitagliptin or a proton pump inhibitor in the preceding 2 months.
3. Vulnerable populations (i.e. cognitively impaired, pregnant women, residing in institutions, University of Alberta students or employees under the supervision of any of the investigators).
4. Children, adolescent or patients with a "contraindication" or "warning" listed in the package insert of any of the study drugs:

   1. Hypersensitivity to sitagliptin or pantoprazole for any component of the formulation.
   2. Renal disease or renal dysfunction (as suggested by serum creatinine levels ≥ 136 µmol/L (males), ≥ 124 µmol/L (females) or abnormal creatinine clearance; or estimated by Glomerular Filtration Rate (GFR) <50 ml/min/1.73m2).
   3. Acute or chronic metabolic acidosis with or without coma (including diabetic ketoacidosis).
5. Uncontrolled hyperglycemia
6. Any subject that in the opinion of the investigator would not be a good candidate for study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-10; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Senior, MD, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta - Clinical Islet Transplant Program, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Senior PA, Koh A, Yau J, Imes S, Dinyari P, Malcolm AJ, Light P, Shapiro AM. Sitagliptin plus pantoprazole can restore but not maintain insulin independence after clinical islet transplantation: results of a pilot study. Diabet Med. 2017 Feb;34(2):204-212. doi: 10.1111/dme.13131. Epub 2016 May 22. PMID 27087519

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period took place between March 2010 thru October 2010. Consent took place in the Clinical Islet Transplant Program at the University of Alberta.
Pre-assignment Details: Patients signed Informed Consent after a consultation with the PI. Then they proceeded through the evaluation phase of the study. During this phase, some patients were excluded based on the protocol's inclusion and exclusion criteria (i.e. lab reports or procedure that did not meet protocol standards).
Groups:
- Sitagliptin + Pantoprazole: Intervention Details:
  Pantoprazole: Starting on Day 1, Pantoprazole 80 mg daily (40 mg every morning and 40 mg every evening) administered orally at the same time each day for a period of 6 months, followed by a three-month washout.
  Sitagliptin: Starting on Day 1, Sitagliptin 100mg once daily administered orally at the same time each day for a period of 6 months, followed by a three-month washout.
Period: Overall Study
Arm/Group | Sitagliptin + Pantoprazole
Started | 8
Completed | 7
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Patients with evidence of early graft insufficiency following a period of insulin independence after one or more islet infusions for c-peptide negative type 1 diabetes participated in the study.
Groups:
- One Arm: Sitagliptin + Pantoprazole: Intervention Details:
  Sitagliptin 100 mg daily and Pantoprazole 40 mg bid for 6 months, followed by a three-month washout:
  Pantoprazole: Starting on Day 1, Pantoprazole 80 mg daily (40 mg every morning and 40 mg every evening) administered orally at the same time each day for a period of 6 months.
  Sitagliptin: Starting on Day 1, Sitagliptin 100mg once daily administered orally at the same time each day for a period of 6 months.
Arm/Group | One Arm: Sitagliptin + Pantoprazole
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 54 [40 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Region of Enrollment [Number; unit: participants]
  Canada | 8
Weight [Mean (Standard Deviation); unit: kg] | 69 (15)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.6 (3.4)
Diabetes Duration Prior to 1st Transplant [Mean (Full Range); unit: years] | 36.1 [24.7 to 50.2]
Number of islet infusions [Median (Full Range); unit: number of islet infusions] | 2 [1 to 4]
Islet equivalents infused [Mean (Standard Deviation); unit: equivalents total] | 814,061 (231,463)
Islet equivalents infused [Mean (Standard Deviation); unit: equivalents per kg] | 12,046 (4,030)
Time since first transplant [Median (Full Range); unit: months] | 67 [25 to 137]
Interval since last transplant [Median (Full Range); unit: months] | 53 [17 to 136]
Time insulin free [Median (Full Range); unit: months] | 47.8 [15.4 to 135.3]
Tacrolimus daily dose [Mean (Standard Deviation); unit: mg] | 4.5 (1.2)
Mycophenolate daily dose [Mean (Standard Deviation); unit: mg] | 1406 (461)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint Will be Insulin Independence After 6 Months of Therapy.
Description: Insulin independence was defined as no insulin use for at least one week, HbA1c < 6.0%, fasting plasma glucose < 7.0 mmol/l, fasting or stimulated c-peptide ≥ 0.5 ng/ml. In addition capillary blood glucose levels could not be >7.8 mmol/l (fasting) or > 10 mmol/l (post-prandial) on more than three occasions in the preceding week. Mean daily insulin use was calculated from the three days prior to study visits. Blinded continuous glucose monitoring (CGM) was performed using the iPro device and Carelink software (Medtronic, Mississauga, ON, CA).
Time Frame: 6 months
Population: Per Protocol Set of participants: The participants of subjects in full analysis set who were: compliant with the protocol, compliant with pre-specified exposure to the treatment regimen, and available for measurements of primary variables.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | One Arm: Sitagliptin + Pantoprazole
Number analyzed (Participants) | 8
proportion of participants | 0.25 [-0.06 to 0.56]
Statistical Analysis 1: Comparison: One Arm: Sitagliptin + Pantoprazole; The sample size of 8 was determined to provide a 95% confidence interval expected width of 0.62 for the proportion of subjects who become insulin independent with treatment. Four of eight subjects (50%) would have to achieve insulin independence in order to reject the null hypothesis with 85% power and one sided alpha of 0.025. Statistical significance was set at 5%. Mean values were computed using Student's t-test while medians were compared using Wilcoxon's test; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

2. Secondary Outcome: Insulin Independence After the 3 Month Washout Period
Description: as for outcome 1
Time Frame: After the 3 month washout period
Population: Per Protocol Set of participants; The subset of participants in full analysis set who were: compliant with the protocol, compliant with pre-specified exposure to the treatment regimen, and available for measurements of primary and secondary variables.
Measure: Number; unit: % of insulin indipendent participants
Groups:
- One Arm: Sitagliptin + Pantoprazole: Intervention Details:
  Sitagliptin 100 mg daily and Pantoprazole 40 mg bid for 6 months, followed by a three-month washout.
  Pantoprazole: Starting on Day 1, Pantoprazole 80 mg daily (40 mg every morning and 40 mg every evening) administered orally at the same time each day for a period of 6 months.
  Sitagliptin: Starting on Day 1, Sitagliptin 100mg once daily administered orally at the same time each day for a period of 6 months.
Arm/Group | One Arm: Sitagliptin + Pantoprazole
Number analyzed (Participants) | 7
% of insulin indipendent participants | 0

3. Secondary Outcome: Insulin Dose (U/Day)
Time Frame: After the 3 month washout period
Reporting Status: Not Posted

4. Primary Outcome: Number of Participants Not Using Insulin for at Least One Week After 6 Months of Therapy
Time Frame: 6 months
Reporting Status: Not Posted

5. Primary Outcome: Number of Participants With HbA1c < 6.0 % After 6 Months of Therapy
Description: HbA1c was measured using method (manufacturer) at baseline, 3, 6 and 9 months.
Time Frame: 6 months
Reporting Status: Not Posted

6. Primary Outcome: Number of Participants With Fasting Plasma Glucose (FPG) < 7 mmol/l After 6 Months of Therapy
Time Frame: 6 months
Reporting Status: Not Posted

7. Primary Outcome: Mean Daily Insulin Use (U/Day) After 6 Months of Therapy
Description: Mean daily insulin use was calculated from the three days prior to study visits and performed at baseline, 3, 6, and 9 months.
Time Frame: 6 months
Reporting Status: Not Posted

8. Primary Outcome: Change From Baseline of GLP-1 Level After One Month of Therapy
Description: Fasting Glucagon-Like Peptide (GLP-1) levels were measured at baseline and one month. Blood samples were collected in p700 vacutainers (Becton Dickinson, Franklin Lakes, NJ) containing a Dipeptidyl peptidase-4 (DPP4) protease inhibitor cocktail to measure total and active GLP-1 in duplicate using a commercially available ELISA (kit manufacturer) and expressed as the ratio of active:total GLP-1.
Time Frame: Baseline and One month
Reporting Status: Not Posted

9. Primary Outcome: Change From Baseline on Gastrin Level After One Month of Therapy
Description: Gastrin levels were measured at baseline and at one month by method (manufacturer).
Time Frame: Baseline and One month
Reporting Status: Not Posted

10. Primary Outcome: HbA1c Plasma Laboratory Value for Participants After 6 Months of Therapy
Description: HbA1c was measured at baseline, 3, 6, and 9 months using method (manufacturer.
Time Frame: 6 months
Reporting Status: Not Posted

11. Primary Outcome: Acute Insulin Responses to Arginine After 6 Months of Therapy
Description: An intravenous arginine stimulation test (AST) [Ryan:2002cg] was performed at baseline, 6, and 9 months to assess Graft function.
Time Frame: 6 months
Reporting Status: Not Posted

12. Primary Outcome: C-peptide Laboratory Value at 90 Minutes After a Mixed Meal Tolerance Test (MMTT) After 6 Months of Therapy
Description: Measuring of C-peptide before and 90 minutes after a mixed meal tolerance test (MMTT) [Ryan:2005ts] at baseline, 6 and 9 months to assess Graft function.
Time Frame: 6 months
Reporting Status: Not Posted

13. Primary Outcome: C-peptide Laboratory Value Before a Mixed Meal Tolerance Test (MMTT) After 6 Months of Therapy
Description: as for outcome 12
Time Frame: 6 months
Reporting Status: Not Posted

14. Primary Outcome: Glucose Laboratory Value at 90 Minutes After Mixed Meal Tolerance Test (MMTT) After 6 Months of Therapy.
Description: Measuring Glucose before and 90 minutes after Mixed Meal Tolerance Test (MMTT) [Ryan: 2005ts] at baseline, 6 and 9 months to assess Graft function.
Time Frame: 6 months
Reporting Status: Not Posted

15. Primary Outcome: Blood Glucose Laboratory Value Before Mixed Meal Tolerance Test (MMTT) After 6 Months of Therapy
Time Frame: 6 months
Reporting Status: Not Posted

16. Primary Outcome: Weight Change From Baseline After 6 Months of Therapy
Description: Measuring the weight change from baseline at months: 1, 3, 6 and 9.
Time Frame: 6 months
Reporting Status: Not Posted

17. Secondary Outcome: Acute Insulin Response to Arginine After the 3 Month Washout Period
Description: An intravenous Arginine stimulation test (AST) [Ryan:2002cg] was performed at baseline, 6, and 9 months to assess Graft function. The Arginine is a proxy for insulin secretory reserve (Robertson:2004br)(Rickels:2007cg) and correlates with islet mass in the context of islet allo-transplant (Ryan:2002cg), auto-transplant (Teuscher:1998eu) and hemipancreatectomy (Seaquist:1992iv). An increase in Arginine (AIRarg) would have suggested an increase in beta cell mass.
Time Frame: 3 months - washout period
Reporting Status: Not Posted

18. Secondary Outcome: HbA1c Plasma Laboratory Value for Participants After the 3 Month Washout Period
Description: Measuring of HbA1c using method (manufacturer) at baseline, and months: 1, 3, 6, 9.
Time Frame: After the 3 month washout period
Reporting Status: Not Posted

19. Secondary Outcome: C-peptide Plasma Laboratory Value at 90 Minutes After a Mixed Meal Tolerance Test (MMTT) at the End of the 3 Month Washout Period.
Description: Measuring of C-peptide before and 90 minutes after a Mixed Meal Tolerance Test (MMTT) [Ryan:2005ts] at baseline, 6 and 9 months to assess Graft function. Ther
Time Frame: After the 3 month washout period
Reporting Status: Not Posted

20. Secondary Outcome: C-peptide Laboratory Value Before a Mixed Meal Tolerance Test (MMTT) After the 3 Month Washout Period.
Description: as for outcome 12
Time Frame: 3 months - washout period
Reporting Status: Not Posted

21. Secondary Outcome: Glucose Laboratory Value at 90 Minutes After Mixed Meal Tolerance Test (MMTT) After the 3 Month Washout Period.
Description: Measuring Blood Glucose before and 90 minutes after Mixed Meal Tolerance Test (MMTT) [Ryan: 2005ts] at baseline, 6 and 9 months to assess Graft function.
Time Frame: 3 months - washout period
Reporting Status: Not Posted

22. Secondary Outcome: Blood Glucose Laboratory Value Before Mixed Meal Tolerance Test (MMTT) After the 3 Month Washout Period
Description: as for outcome 21
Time Frame: After the 3 month washout period
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | One Arm: Sitagliptin + Pantoprazole
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | One Arm: Sitagliptin + Pantoprazole (N=8)
Nausea or Diarrhea (Gastrointestinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The major weaknesses of the study are the small sample size and the lack of a control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes